CLINICAL TRIAL: NCT07132762
Title: The Effect of Extracorporeal Shock Wave Therapy (ESWT) Added to Conservative Treatment on Pain, Disability, and Ultrasonographic Outcomes in Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: The Effect of ESWT Added to Conservative Treatment on Pain, Disability, and Ultrasonographic Outcomes in Chronic Low Back Pain
Acronym: ESWT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Füsun Ardıç, PROFESSOR, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PamukkaleU.ftr-FArdıç-002
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Low Back Pain
Keywords: Extracorporeal Shockwave Therapy treatment (ESWT); Elastography; physical therapy; chronic low back pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT + Conventional Physical Therapy Group (Experimental): A total of 6 sessions of extracorporeal shock wave therapy (ESWT) will be administered twice a week, along with 15 sessions of conventional physical therapy applied five times per week. Each conventional physical therapy session will include 20 minutes of hot pack application, 20 minutes of conventional transcutaneous electrical nerve stimulation (TENS), 5 minutes of ultrasound therapy at an intensity of 1.5 W/cm², and core stabilization exercises performed under the supervision of a physiotherapist. The treatment program will be carried out over a total period of 3 weeks. Each ESWT session will last approximately 15 minutes. ESWT will be applied with the patient positioned in the prone position, using an energy density of 0.15 mJ/mm², at a frequency of 4 Hz, and delivering 1,500 shock waves per session. The application will target the right and left paravertebral muscles between the L3 and S1 spinal segments.
  Interventions: Device: Radial Extracorporeal Shock Wave Therapy; Other: Conventional rehabilitation
- Conventional Physical Therapy Group (Active Comparator): A total of 15 sessions of conventional physical therapy will be administered, five times per week. Each session will include 20 minutes of hot pack application, 20 minutes of conventional transcutaneous electrical nerve stimulation (TENS), 5 minutes of ultrasound therapy at 1.5 W/cm², and core stabilization exercises performed under the supervision of a physiotherapist. The treatment will be applied over a total period of 3 weeks.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Device: Radial Extracorporeal Shock Wave Therapy — A total of 6 sessions of ESWT, applied twice a week. Each ESWT session will last approximately 15 minutes. ESWT will be administered with the patient in the prone position, using an energy density of 0.15 mJ/mm², at 4 Hz frequency, and 1,500 shock waves per session.
  The ESWT application will be performed on the right and left paravertebral muscles between the L3 and S1 segments.
  Arms: ESWT + Conventional Physical Therapy Group
Other: Conventional rehabilitation — A total of 15 sessions of conventional physical therapy will be administered, five times per week. Each session will include 20 minutes of hot pack application, 20 minutes of conventional transcutaneous electrical nerve stimulation (TENS), 5 minutes of ultrasound therapy at 1.5 W/cm², and core stabilization exercises performed under the supervision of a physiotherapist. The treatment will be applied over a total period of 3 weeks.

SUMMARY:
Chronic low back pain (CLBP) is a major public health concern worldwide, leading to reduced quality of life and significant work loss. It is defined as pain lasting more than 12 weeks between the lumbar and sacral spinal segments. The global prevalence of CLBP ranges from 13.1% to 20.3%, and the number of affected individuals has increased from 370 million in 1990 to 570 million in 2017.

Core muscles, including the multifidus, erector spinae, transversus abdominis, psoas major, and quadratus lumborum, play a key role in spinal stabilization. In patients with CLBP, dysfunction and loss of synergy among these muscles can compromise spinal balance. Prolonged poor posture can reduce the strength and endurance of the lumbar erector spinae, multifidus, and transversus abdominis, leading patients to compensate by overusing the erector spinae, rectus abdominis, and oblique abdominal muscles. This compensation is considered one of the primary contributors to chronic low back pain.

These deep core muscles can be objectively evaluated using ultrasonography (USG), a non-invasive, inexpensive, and accessible imaging method. Strain elastography, a quantitative ultrasonographic technique, is increasingly used to assess tissue stiffness and monitor structural changes in muscle over time.

Conventional treatments for CLBP include pharmacotherapy, exercise, and physical therapy. In recent years, extracorporeal shock wave therapy (ESWT) has emerged as a non-invasive, easily applicable, and low-risk treatment method. ESWT is widely used in various musculoskeletal conditions such as lateral epicondylitis, patellar tendinopathy, and calcific tendinitis of the shoulder. Studies have shown that ESWT provides pain relief and functional improvement in patients with CLBP through its angiogenic, anti-inflammatory, analgesic, and tissue-regenerative effects.

Several studies have demonstrated the positive impact of ESWT on pain reduction and functional recovery in CLBP. A recent meta-analysis reported that ESWT significantly reduces pain in CLBP patients and may be superior to other conservative treatments. Yue et al. (2021) highlighted the short-term benefits of ESWT in reducing pain and disability, while also emphasizing the need for well-designed randomized controlled trials (RCTs) to establish high-quality evidence. Similarly, Wu et al. (2023) underscored the necessity of including objective outcomes in future RCTs to better evaluate the efficacy of ESWT.

Although numerous studies have assessed the effects of ESWT on pain, disability, and functional outcomes in CLBP, to date, no study has objectively evaluated its effectiveness using ultrasonographic strain elastography focusing on the elasticity and stiffness of core muscles.

This study aims to be one of the first to assess the long-term effects of ESWT using objective measures. Its contribution to the literature lies in evaluating the efficacy of ESWT, when added to conventional physical therapy, through long-term monitoring with ultrasonographic strain elastography in patients with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Non-specific low back pain lasting more than three months

Exclusion Criteria:

* Specific lumbar spine diseases (radicular pain, spinal stenosis, infection)
* History of trauma, fracture, surgery, or presence of scar tissue in the lumbar region
* Presence of a disease that may affect muscle stiffness, such as collagen tissue disorders, hemiplegia, multiple sclerosis, or myopathies
* Malignancy, pregnancy, severe hypertension
* Coagulopathy, chronic heart disease
* Ankylosing spondylitis
* Diseases that may initially affect lumbar mobility and pain, such as leg length discrepancy, hip prosthesis, or scoliosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, 3rd week, 12th week
  The Visual Analog Scale (VAS), a valid and reliable method for measuring pain intensity, will be used. VAS is a 10-centimeter-long horizontal line that allows patients to assess their pain or symptoms. The left end of the line (0 cm) typically represents "No Pain" or "Painless," while the right end (10 cm) indicates "Unbearable Pain" or "Worst Possible Pain." Participants will be asked to mark a point on the line that corresponds to their current level of pain or symptoms. The marked point is then measured and recorded as a score ranging from 0 to 10. The resulting VAS scores will be used to quantitatively assess the severity of participants' pain or symptoms.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline, 3rd week, 12th week
  The Oswestry Disability Index (ODI) will be used for evaluation. The ODI is used to measure the degree of functional limitations caused by pain in patients with low back pain. It assesses pain intensity, personal care (such as washing and dressing), lifting, walking, sitting or standing, sleeping, sexual life, social life, and traveling/mobility. Each component is scored on a scale from 0 to 5, with 5 indicating the highest level of disability. The index is calculated by dividing the total score by the maximum possible score and multiplying the result by 100 to obtain a percentage score representing the level of disability.
Sonoelastography -Strain Index: | Baseline, 3rd week ,12th week
  Sonoelastography strain index, which is a quantitative analysis method used to measure elasticity, will be used. With elastographic quantitative analysis, a software feature of the ultrasound system, the color distribution in a selected area is numerically measured through single or multiple boxes, and an elasticity index is calculated for the measured area. The elasticity index is a value between 0.0 and 6.0 and is determined by the reflected color distribution within the selected region. A higher value indicates greater stiffness and is represented predominantly by the color blue on the screen. While the elasticity index is calculated separately for the reference area and the muscle, the system automatically calculates the elasticity ratio as muscle/reference area.

CONTACTS AND LOCATIONS:
Overall Officials: Füsun Ardıç, Professor, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)